CLINICAL TRIAL: NCT07237295
Title: CommunityRx-Chronic Kidney Disease in Rural North Carolina
Brief Title: CommunityRx-Chronic Kidney Disease
Acronym: CRx-CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Goshen Medical Center (Unknown); James McFarlin Community Development, Inc. (Other); Johns Hopkins University (Other); Project GRACE (Unknown); Project Momentum, Inc. (Industry); Unite Us (Unknown); University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-2006; 1U01DK137262 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease (Stages 1-4)
Keywords: Chronic disease management; Health-related social needs; Rural health; Self-efficacy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: We will individually randomize eligible participants to the CRx-CKD or usual care in a 1:1 ratio stratified by the number of providers (1, 2, or 3+) at each clinic site.
Who Masked: Investigator
Masking Description: Investigators are masked to participant assignments. Unmasked research staff support the navigators as needed in enrollment and follow-up procedures. Double-masking is not possible, as participants in the active condition will receive the three CommunityRx-Chronic Kidney Disease components described during the consent process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention + usual care (Experimental): This arm will receive the intervention in addition to usual care.
  Interventions: Behavioral: CommunityRx-Chronic Kidney Disease
- Usual care only (No Intervention): This arm will not receive the intervention.

INTERVENTIONS:
Behavioral: CommunityRx-Chronic Kidney Disease — CommunityRx-Chronic Kidney Disease (CRx-CKD) is an evidence-based, low-intensity, health information technology-driven intervention designed to support chronic kidney disease management in rural eastern North Carolina. CRx-CKD integrates medical (e.g., blood pressure and glucose monitoring, eye and foot care), social (food, housing, transportation), and self-care (weight and stress management, exercise) resources. CRx-CKD comprises three components: brief education on integrated chronic kidney disease needs, a chronic kidney disease care plan that includes integrated care referrals, and clinic navigator-led, longitudinal support (12 months) for chronic kidney disease patients.
  Other Names: CRx-CKD; HealtheRx
  Arms: Intervention + usual care

SUMMARY:
In the United States, the burden of chronic kidney disease rests disproportionately on rural communities. This study evaluates the implementation and effectiveness of CommunityRx-Chronic Kidney Disease (CRx-CKD); this health information technology intervention integrates medical, social, and self-care resources to improve CKD management in rural eastern North Carolina. Through a partnership among local primary care centers, community organizations, and researchers, CRx-CKD will strengthen rural care networks, improve CKD management, and enhance the well-being of rural communities.

DETAILED DESCRIPTION:
Approximately one in seven adults in the United States lives with chronic kidney disease. Chronic kidney disease typically worsens with time and, in its final stage, can result in kidney failure. Contextual factors in rural, eastern North Carolina communities impede optimal management of chronic kidney disease multimorbidity. In these communities, geographical barriers to medical care, dwindling resources, and underdeveloped health infrastructure have worsened chronic kidney disease outcomes. CommunityRx-CKD (CRx-CKD) is an evidence-based, low-intensity, health information technology-driven intervention designed to support chronic kidney disease management in rural eastern North Carolina. CRx-CKD integrates medical (e.g., blood pressure and glucose monitoring, eye and foot care), social (food, housing, transportation), and self-care (weight and stress management, exercise) resources. CRx-CKD comprises three components: brief education on integrated chronic kidney disease needs, a chronic kidney disease care plan that includes integrated care referrals, and clinic navigator-led, longitudinal support (12 months) for chronic kidney disease patients in our trial. Our multidisciplinary, community-engaged research team will test the effects of CRx-CKD through three related aims.

This pragmatic individual-randomized, two-arm, single-blind trial in 25 rural primary care clinics in 12 rural eastern North Carolina counties (n=634 adults with CKD) assesses the effect of CRx-CKD on acute healthcare utilization (primary outcome), self-efficacy for finding resources, knowledge and sharing of integrated care resources, resource use, number of unmet needs over time, ambulatory care utilization, and health-related quality of life. The researchers hypothesize that 12-month acute healthcare utilization will differ between participants receiving CRx-CKD and those receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic kidney disease defined as ≥1 ICD-10 CKD codes (excluding end-stage kidney disease) or CKD biomarkers (estimated glomerular filtration rate ≤ 60 ml/min, albuminuria ≥30 mg/24h)
* At least one clinic visit at Goshen Medical Center in 12 months before enrollment

Exclusion Criteria:

* Limited life expectancy (e.g., advanced cancer, end-stage liver disease, hospice)
* Active cancer treatment
* Living in a skilled nursing facility
* Dementia/other significant cognitive impairment/inability to participate in the informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean number of 911 calls | Baseline, 3 months, 6 months, 9 months, 12 months
  Number of 911 calls is self-reported with a look-back period of 3 months in response to an item originally used in the DIAMOND RCT: "How many times has 911 been called (either by yourself or someone acting on your behalf)?"
Mean number of emergency room visits | Baseline, 3 months, 6 months, 9 months, 12 months
  Number of emergency room visits is the sum of two self-reported items with a look-back period of 3 months, originally used in the DIAMOND RCT:
  1. "How many times did the ambulance take you to the emergency room?"
  2. "How many times did you go to the emergency room without an ambulance?"
Mean number of after-hours or urgent care clinic visits | Baseline, 3 months, 6 months, 9 months, 12 months
  Number of after-hours of urgent care clinic visits is self-reported with a look-back period of 3 months in response to an item originally used in the DIAMOND RCT: "How many times did you go to the after-hours medical clinic?"
Mean number of hospital admissions | Baseline, 3 months, 6 months, 9 months, 12 months
  Number of hospital admissions is self-reported with a look-back period of 3 months in response to an item originally used in the DIAMOND RCT: "How many times were you admitted to the hospital?"

SECONDARY OUTCOMES:
Self-efficacy to find community-based resources | Baseline, 6 months, 12 months
  Self-efficacy to find community-based resources is measured using an item developed from Bandura's self-efficacy theory and used in prior CommunityRx trials: "How confident are you in your ability to find resources in your community that help you manage your health?" Responses will be assessed on a 5-point Likert scale ranging from '1' (not at all confident) to '5' (completely confident).
Number of participants reporting knowledge community-based resources | Baseline, 6 months, 12 months
  Knowledge of community-based resources is measured using 10 self-reported items adapted and tested in prior CommunityRx studies: "Do you know of places in your community that offer [specific resources]?" We will report the number of participants endorsing knowledge of 0, 1, 2, 3 or 4+ resource types.
Mean attitude about community-based resources | Baseline, 6 months, 12 months
  Attitude about community-based resources is measured using a self-report Likert item adapted and tested in prior CommunityRx studies: "Your community has the resources you need to manage your health." Response range from '1' (strongly agree) to '5' (strongly disagree).
Number of participants reporting use of community-based resources | Baseline, 6 months, 12 months
  Use of community resources is measured using 10 self-reported survey items adapted and tested in prior CommunityRx studies: "Have you received services from places like this for you or your household in the last 6 months?" We will report the number of participants endorsing utilization of 0, 1, 2, 3 or 4+ resource types.
Number of participants sharing community-based resources | Baseline, 6 months, 12 months
  Sharing of community resources is measured using 10 self-reported survey items adapted and tested in prior CommunityRx studies: "Have you told anyone about places like this in the past 6 months?" We will report the number of participants endorsing sharing 0, 1, 2, 3 or 4+ resource types.
Mean number of physician office visits | Baseline, 3 months, 6 months, 9 months, 12 months
  Number of physician office visits is self-reported with a look-back period of 3 months in response to an item originally used in the DIAMOND RCT: "How many times have you seen a physician for an office visit?"
Number of health-related social needs | Baseline, 6 months, 12 months
  Health-related social needs are measured via the Accountable Health Communities Health-Related Social Needs Screener. This measure includes ten items evaluating participant needs across the domains of: housing, food, transportation, utilities, and interpersonal violence. Higher scores indicate greater needs.
Mean Patient-Reported Outcome Measurement Information System (PROMIS) Global-10 score | Baseline, 6 months, 12 months
  The PROMIS Global-10 measures general health-related quality-of-life. Response options are presented as nine 5-point and one 11-point Likert scales. Higher scores indicate greater health-related quality-of-life.

OTHER OUTCOMES:
Mean Medical Mistrust Index score | Baseline, 6 months, 12 months
  The Medical Mistrust Index measures mistrust in the health system. Participants respond to 7 Likert scale items assessing the extent to which they disagree or agree with a given statement (e.g., "You'd better be cautious when dealing with health care organizations"). Items are scored from '1' (strongly disagree) to '4' (strongly agree). Higher scores indicate greater levels of mistrust in the health system.
Mean estimated glomerular filtration rate (eGFR) in mL/min/1.73m² | Baseline, 6 months, 12 months
  eFGR is abstracted from participant electronic medical records.
Mean creatinine in µmol/L | Baseline, 6 months, 12 months
  Creatinine is abstracted from participant electronic medical records.
Mean number of comorbidities | Baseline, 6 months, 12 months
  Comorbidities are abstracted from participant electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav J Dave, DrPH, MPH, MBBS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Goshen Medical Center, Beulaville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with The University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with The University of North Carolina at Chapel Hill